CLINICAL TRIAL: NCT01069211
Title: Assessment of Clinical Outcomes After Letrozole Treatment According to the Estrogen Receptor Expression in Postmenopausal Women With Hormone Receptor Positive Breast Cancer
Brief Title: Clinical Outcomes After Letrozole Treatment According to the Estrogen Receptor Expression in Postmenopausal Women
Acronym: LETTER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korean Breast Cancer Study Group (Other)
Responsible Party: Joon Jeong, Gangnam Severance Hospital, South Korea.
Other Study IDs: KBCSG006
Record Dates: First submitted 2010-02-14; First posted 2010-02-17 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer, Letrozole; postmenopause; hormone receptor positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast Cancer Tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ER expression : Low: Patients were postmenopausal women with hormone receptor positive breast cancer. All patients should be 3 or 4 point of total Allred score.
- ER expression : Intermediate: Patients were postmenopausal women with hormone receptor positive breast cancer. All patients should be 5 or 6 point of total Allred score.
- ER expression : High: Patients were postmenopausal women with hormone receptor positive breast cancer. All patients should be 7 or 8 point of total Allred score.

SUMMARY:
The purpose of this study is to assess clinical outcomes after Letrozole treatment according to the estrogen receptor expression in postmenopausal women with hormone receptor positive breast cancer.

DETAILED DESCRIPTION:
This study aimed at evaluating following:

1. Validity Assessment:

   1. Primary End Point: To evaluate 5-year diseae free survival rate after Letrozole treatment according to the estrogen receptor expression in postmenopausal women
   2. Secondary End Point: To evaluate overall survival rate(OS) and Time to distance recurrence(TTDR) after Hormonal therapy in postmenopausal women with hormone receptor positive breast cancer
2. Safety Assessment: To evaluate all adverse events including serious adverse events after Letrozole treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with estrogen receptor(+) and/or progesterone receptor(+)
2. Postmenopausal state was defined the following conditions, at least one of a, b

   1. Serum FSH ≥ 30 mIU/mL and Amenorrhea ≥ 1 year for below 55 years, over than 55 years
   2. Bilateral oophorectomy
3. Patients have undergone surgery of the breast cancer within 12 weeks and terminated chemotherapy after surgery within 4 weeks.
4. WHO(ECOG) performance status 0-2
5. Adequate haematological function, renal function, hepatic function.
6. No evidence of metastasis.

Exclusion Criteria:

1. Metachronous bilateral breast cancer.
2. Metastatic breast cancer (stage IV)
3. Other hormone therapy and Hormonal replacement therapy given within the previous 4 weeks, except for Estring, Vagifem, Estrogen Cream.
4. Patients with Child-Pugh grade C, serum creatinine>2xUNL
5. Patients with gastrectomy, small bowel resection, malabsorption syndrome and dysphagia.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients recruited into the study are postmenopausal women with estrogen receptor positive breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 876 (Estimated)
Dates: Start 2010-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | the first 5 years after enrollment

SECONDARY OUTCOMES:
Adverse effect | the first 5 years after enrollment
Overall Survival | the first 5 years after enrollment
Time to Distant Recurrence (TTDR) | the first 5 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Joon Jeong, MD, Principal Investigator — Department of Surgery, Gangnam Severance Hospital, South Korea
Locations (1):
- Joon Jeong, Seoul, South Korea

REFERENCES:
- [Derived] Ahn SG, Nam SJ, Ahn SH, Jung Y, Park HK, Lee SJ, Kang SS, Han W, Park KH, Park YL, Lee J, Youn HJ, Kim JH, Yoo Y, Song JY, Ko BK, Gwak G, Chung MS, Kim SY, Cho SH, Kim D, Chang MC, Moon BI, Kim LS, Kim SJ, Park MH, Kim TH, Cho J, Lim CW, Bae YT, Gong G, Bae YK, Lee A, Jeong J. Clinical Outcomes Following Letrozole Treatment according to Estrogen Receptor Expression in Postmenopausal Women: LETTER Study (KBCSG-006). J Breast Cancer. 2021 Apr;24(2):164-174. doi: 10.4048/jbc.2021.24.e17. Epub 2021 Mar 25. PMID 33818022